CLINICAL TRIAL: NCT04058184
Title: Prepulse Inhibition of the Startle Response in Youth Contact Sports Players
Brief Title: Prepulse Inhibition in Youth Contact Sports Players
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Wake Forest University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00051757
Record Dates: First submitted 2019-08-08; First posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-07

CONDITIONS: Reflex, Abnormal
Keywords: Prepulse Inhibition; Startle Response
MeSH Terms: conditions — Reflex, Abnormal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Contact sports players: Athletes who engage in contact sports, football for example. Participation in this study will involve listening to sudden, very brief bursts of noise (startle blocks) and tones, and responding with a keypress to certain tones. Electromyogram (EMG) will measure the electrical activity generated from movement of the orbicularis oculi muscle during the startle blocks.
- Non-contact sports players: Athletes who engage in non-contact sports, swimming for example.Participation in this study will involve listening to sudden, very brief bursts of noise (startle blocks) and tones, and responding with a keypress to certain tones. Electromyogram (EMG) will measure the electrical activity generated from movement of the orbicularis oculi muscle during the startle blocks.

SUMMARY:
The study's main research question will be investigating whether or not there is a significant difference in Prepulse Inhibition (PPI) as well as startle response probability and magnitude between contact and noncontact youth sports players. The study team will test these questions using a controlled laboratory scenario in which the presentation of startle stimuli can be observed, measured, and quantified in order to compare the results between the two sample populations. During preliminary testing, the study team can predict that there will be no significant differences between contact sports players and noncontact sports players in their startle reactivity and level of exhibited PPI. Based on previous literature, the study team hypothesizes that those in the contact sports group will experience greater startle reactivity and less PPI than those in the noncontact sports group when they are tested at the end of their sports season. Using this information, the present study will allow for additional understanding of the neurological and physiological behaviors associated with subconcussive head impacts.

This study will assess and determine whether prepulse inhibition in youth contact sports players and non-contact sports players, both before and after a sports season, will significantly differ. Measures will include the startle magnitude, startle probability, reaction time, and accuracy of tone detection responses.

DETAILED DESCRIPTION:
Our main research question will be investigating whether or not there is a significant difference in PPI, as well as startle response probability and magnitude between contact and noncontact youth sports players. The study team will test these questions using a controlled laboratory scenario in which the presentation of startle stimuli can be observed, measured, and quantified in order to compare the results between the two sample populations. During preliminary testing, the study team can predict that there will be no significant differences between contact sports players and noncontact sports players in their startle reactivity and level of exhibited PPI. Based on previous literature, the study team hypothesizes that those in the contact sports group will experience greater startle reactivity and less PPI than those in the noncontact sports group when they are tested at the end of their sports season. Using this information, the present study will allow for additional understanding of the neurological and physiological behaviors associated with subconcussive head impacts.

This study will assess and determine whether prepulse inhibition in youth contact sports players and non-contact sports players, both before and after a sports season, will significantly differ. Measures will include the startle magnitude, startle probability, reaction time, and accuracy of tone detection responses.

The current study is a case-control study, examining the contact sports players as the testing sample and the noncontact sports players as the control sample.

* Participants will arrive and hear an introduction of the study.
* Participants (and their parent/guardian if under the age of 18) will read and sign an informed consent and/or informed assent form.
* Participants will complete a series of questionnaires prior to electrode placement.

  * The Health History Questionnaire will be completed first to determine participant eligibility.
  * The STAI will be completed next to be used for further analysis in the data compilation.
* Participants will have three electrodes placed on the skin.

  * Two electrodes will be placed underneath the left eye as the nasal and temporal electrodes.
  * One electrode will be placed on the left temple as the ground electrode.
  * These electrodes connect to the Biopac apparatus, the software that measures the participant's EMG activity.
* The procedure of the study will be thoroughly explained to the participants. They will be instructed to wear headphones that will deliver the acoustic startle stimuli and to remain as still and quiet as possible during the startle blocks.

  * There will be a total of two startle blocks: baseline and testing.
  * The baseline startle block will consist of a combination of prepulses at 70 decibels of 800 and 1000 Hz frequency tones for a duration of 30 milliseconds presented with an onset of 120 milliseconds prior to the presentation of the startle stimulus of 100 decibels of broadband noise for 50 milliseconds on some trials.
  * The testing block will also consist of prepulses at 70 decibels of 800 and 1000 Hz frequency tones for a duration of 30 milliseconds presented with an onset of 120 milliseconds prior to the presentation of the startle stimulus of 100 decibels of broadband noise for 50 milliseconds on some trials. For the testing block, participants will be asked to respond on a keypad when they hear the lower prepulse tone of 800 Hz.
  * Startle stimuli will be presented via headphones. Startle stimuli will be presented from the Superlab software program which will run from the testing room.
* After the testing block, the electrodes will be removed from the participant's skin.
* Participants will be thoroughly debriefed on the aims of the current study.

This study will take place in the MRI suite of Wake Forest Baptist Health. A single room within the suite will be designated for the PPI testing, in order to control for external noise factors.

After the consent process, subjects will be asked to fill out a brief health history questionnaire. This is for the purpose of determining the subject's eligibility to participate in the study. Subjects will also be asked to complete an STAI form, and this will be used later during data analysis.

This study will last approximately one hour. The introduction and consent process will take about 10 minutes. The questionnaire process is expected to take about 10 minutes. The application of sensors should take about 10 minutes. The testing process, including the explanation of both startle blocks, should last about 20 minutes. The sensor removal and debriefing process will last about 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

• Participants are specifically recruited for this study due to their involvement on a sports team that may or may not expose them to head impacts.

Exclusion Criteria:

• Subjects on psychostimulant, antidepressant, or anxiolytic medications, as well as subjects who have experienced hearing loss, will not be eligible to participate.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants who participate on a sports team who range in age from 13 to 19.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Startle Magnitute | baseline
  collected from each participant's raw EMG data
Startle Magnitute | startle test up to 1 hr from baseline
  collected from each participant's raw EMG data
Startle Probability | baseline
  collected from each participant's raw EMG data
Startle Probability | startle test up to 1 hr from baseline
  collected from each participant's raw EMG data
Percentage of Prepulse Inhibition | baseline test
  collected from each participant's raw EMG data
Percentage of Prepulse Inhibition | startle test up to 1 hr from baseline
  collected from each participant's raw EMG data

SECONDARY OUTCOMES:
Reaction Time | baseline test
  data collected from applicable subject's response pad
Reaction Time | startle test up to 1 hr from baseline
  data collected from applicable subject's response pad
Accuracy Measures | baseline test
  data collected from applicable subject's response pad
Accuracy Measures | startle test up to 1 hr from baseline
  data collected from applicable subject's response pad

CONTACTS AND LOCATIONS:
Overall Officials: Blumenthal, Principal Investigator — Wake Forest University
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blumenthal TD. Presidential Address 2014: The more-or-less interrupting effects of the startle response. Psychophysiology. 2015 Nov;52(11):1417-31. doi: 10.1111/psyp.12506. Epub 2015 Aug 18. PMID 26283146
- [Background] Blumenthal TD, Reynolds JZ, Spence TE. Support for the interruption and protection hypotheses of prepulse inhibition of startle: evidence from a modified Attention Network Test. Psychophysiology. 2015 Mar;52(3):397-406. doi: 10.1111/psyp.12334. Epub 2014 Sep 19. PMID 25234706
- [Background] Washington JR, Blumenthal TD. Effects of a startle stimulus on response speed and inhibition in a go/no-go task. Psychophysiology. 2015 Jun;52(6):745-53. doi: 10.1111/psyp.12400. Epub 2014 Dec 23. PMID 25532594
- [Background] Jepma M, Wagenmakers EJ, Band GP, Nieuwenhuis S. The effects of accessory stimuli on information processing: evidence from electrophysiology and a diffusion model analysis. J Cogn Neurosci. 2009 May;21(5):847-64. doi: 10.1162/jocn.2009.21063. PMID 18702584
- [Background] Thorne GL, Dawson ME, Schell AM. Attention and prepulse inhibition: the effects of task-relevant, irrelevant, and no-task conditions. Int J Psychophysiol. 2005 May;56(2):121-8. doi: 10.1016/j.ijpsycho.2004.11.006. Epub 2005 Jan 21. PMID 15804447